CLINICAL TRIAL: NCT04149704
Title: Videos for Advance Care Planning in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jennifer Snaman, MD, MS, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-409
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Results first posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-12

CONDITIONS: Advanced Cancer
Keywords: Advanced Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACP video decision aid (Experimental): The research study procedures include: screening for eligibility and study interventions including questionnaires and follow up visits.
  * In-person interview where the patient and caregiver together will randomized to either the video aid intervention or standard care
  * 10 minute video decision aid: describing the goals-of-care options .
  * Follow telephone interview at 3 months
  Interventions: Behavioral: ACP video decision aid
- Standard Care (Active Comparator): The research study procedures include: screening for eligibility and study interventions including questionnaires and follow up visits.
  * In-person interview where the patient and caregiver together will randomized to either the video aid intervention or standard care
  * Receive the verbal description of the three types of care
  * Follow telephone interview at 3 months
  Interventions: Other: Usual Care-

INTERVENTIONS:
Behavioral: ACP video decision aid — 10 minute video decision aid describing the goals-of-care options
  Arms: ACP video decision aid
Other: Usual Care- — Verbal description of the three types of care
  Arms: Standard Care

SUMMARY:
This study is a randomized trial of adolescent and young adults with advanced cancer and their caregivers to assess preferences for care in advanced cancer. This research study is examining the similarities and differences between patient's and caregiver's goals of cancer care.

The names of the study interventions involved in this study may include:

* Questionnaires
* Video
* Phone Interview

DETAILED DESCRIPTION:
The research study procedures include: screening for eligibility and study interventions including questionnaires and follow up visits.

- Patients and their caregivers will be randomized into the same group; either ACP video decision aid intervention or usual care.

* Patients' and caregivers' knowledge, preferences (goals of care, CPR, ventilation), and decisional conflict be assessed before and after the ACP video decision aid intervention or usual care.
* Participants will be in this research study for up to 3 months with only 2 study visits.
* It is expected that about 100 people (50 patients and 50 caregivers) will take part in this research study.

ELIGIBILITY:
All patients will be recruited from the outpatient clinics of Dana-Farber Cancer Institute (both pediatric and adult clinics),the inpatient settings of Boston Children's Hospital and Brigham and Women's Hospital, the inpatient or outpatient clinics of Massachusetts General Hospital, or virtually. Eligible study participants will give written consent to the primary investigator or study staff member before initiation of study procedures if recruited in-person. If participants are enrolled and complete study procedures virtually, they will provide verbal consent before initiating study procedures.

If in-person visits cannot be conducted, eligible participants will be still be mailed a pre-notice letter that offers the chance for participants to opt-out or opt-in via email or phone call. After one week, we will call participants we have not heard from and ask if they would consider participating.

Patient Eligibility criteria will include patients who are:

i) Diagnosed with advanced cancer (i.e., initial first-line therapy is unsuccessful, marked by progression or relapsed disease) ii) Aged between 18-39, which is the legal age for completing an ACP document (e.g., POLST/MOLST); iii) Speak English; and iv) Have a caregiver or identified surrogate decision maker who is able to participate.

v) Treated at Dana-Farber Cancer Institute or Massachusetts General Hospital

Exclusion criteria will include:

i) A diagnosis of low-grade glioma given the fact that progressive or relapsed low grade may not be clinically characterized as advanced disease and associated poor prognosis.

ii) Visually impaired (note, hearing impaired is not an exclusion as the video is closed captioned); iii) Psychological state not appropriate for ACP discussions as determined by the primary oncologist; and, iv) Unable to participate in ACP discussions due to mental incapacity as determined by the Short Portable Mental Status Questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Snaman, MD, MS, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] Snaman JM, Feifer D, Helton G, Chang Y, El-Jawahri A, Volandes AE, Wolfe J. A Pilot Randomized Trial of an Advance Care Planning Video Decision Support Tool for Adolescents and Young Adults With Advanced Cancer. J Natl Compr Canc Netw. 2023 Jul;21(7):715-723.e17. doi: 10.6004/jnccn.2023.7021. PMID 37433434

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruited while in clinic; shift to almost all virtual recruitment in late 2020. Eligible individuals received a latter explaining the study and were called one week later to provide further details and determine interest.
Pre-assignment Details: All enrolled participant completed a baseline survey prior to randomization
Groups:
- Standard Care - Patients; Standard Care - Caregivers: The research study procedures include: screening for eligibility and study interventions including questionnaires and follow up visits.
  * In-person interview where the patient and caregiver together will randomized to either the video aid intervention or standard care
  * Receive the verbal description of the three types of care
  * Follow telephone interview at 3 months
  Usual Care: Verbal description of the three types of care
- ACP Video Decision Aid - Patients; ACP Video Decision Aid - Caregivers: The research study procedures include: screening for eligibility and study interventions including questionnaires and follow up visits.
  * In-person interview where the patient and caregiver together will randomized to either the video aid intervention or standard care
  * 10 minute video decision aid: describing the goals-of-care options .
  * Follow telephone interview at 3 months
  ACP video decision aid: 10 minute video decision aid describing the goals-of-care options
Period: Baseline and Immediately Post
Arm/Group | Standard Care - Patients | Standard Care - Caregivers | ACP Video Decision Aid - Patients | ACP Video Decision Aid - Caregivers
Started | 26 | 25 | 25 | 26
Completed (3 month follow up time point) | 26 | 25 | 25 | 26
Not Completed | 0 | 0 | 0 | 0
Period: Three Month Follow-up
Arm/Group | Standard Care - Patients | Standard Care - Caregivers | ACP Video Decision Aid - Patients | ACP Video Decision Aid - Caregivers
Started | 26 | 25 | 25 | 26
Completed | 21 | 21 | 20 | 20
Not Completed | 5 | 4 | 5 | 6
Not completed — Death | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 4 | 5 | 5
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Not completed as dyad (one member of dayd did not complete initial timepoint so withdrawn from study | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: participants were enrolled as AYA and caregiver dyads; presented here as individual participants.
Groups:
- Standard Care - Patient; Standard Care - Caregiver: The research study procedures include: screening for eligibility and study interventions including questionnaires and follow up visits.
  * In-person interview where the patient and caregiver together will randomized to either the video aid intervention or standard care
  * Receive the verbal description of the three types of care
  * Follow telephone interview at 3 months
  Usual Care: Verbal description of the three types of care
- ACP Video Decision Aid - Patient; ACP Video Decision Aid - Caregiver: The research study procedures include: screening for eligibility and study interventions including questionnaires and follow up visits.
  * In-person interview where the patient and caregiver together will randomized to either the video aid intervention or standard care
  * 10 minute video decision aid: describing the goals-of-care options .
  * Follow telephone interview at 3 months
  ACP video decision aid: 10 minute video decision aid describing the goals-of-care options
- Total: Total of all reporting groups
Arm/Group | Standard Care - Patient | Standard Care - Caregiver | ACP Video Decision Aid - Patient | ACP Video Decision Aid - Caregiver | Total
Number analyzed (Participants) | 26 | 26 | 24 | 24 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.5 (6.1) | 41.3 (13.6) | 32.7 (5.6) | 43.0 (13.8) | 37.6 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 14 | 14 | 58
  Male | 10 | 12 | 10 | 10 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 2
  Not Hispanic or Latino | 24 | 24 | 22 | 23 | 93
  Unknown or Not Reported | 1 | 1 | 2 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 2 | 0 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 21 | 22 | 21 | 20 | 84
  More than one race | 0 | 0 | 2 | 2 | 4
  Unknown or Not Reported | 1 | 2 | 1 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 26 | 26 | 24 | 24 | 100

OUTCOME MEASURES:

1. Primary Outcome: Increased Concordance Rate in Stated Goals of Care (Life-prolonging Medical Care, Selective Medical Care, or Comfort-focused Care)
Description: AYA with advanced cancer and caregivers randomized to the video will have higher concordance in their stated goals of care between patients and caregivers at 3 month compared to baseline
Time Frame: baseline, 3 months
Population: Analyzed as dyad. If one individual of the dyad did not complete study procedures, those results were not analyzed. One AYA assigned to standard care did not have a caregiver that was able to participate. One AYA of a caregiver assigned to video decision aid was unable to participate. As the unit of measurement was the DYAD, these two individuals (one standard arm, one video) were not analyzed although they did complete enrollment and baseline and follow-up assessments (but not 3 month)
Measure: Count of Participants; unit: Participants
Groups:
- ACP Video Decision Aid: * In-person interview where the patient and caregiver dyad will randomized to either the video aid intervention or standard care and complete baseline questionnaire
  * 10 minute video decision aid: describing the goals-of-care options
  * Follow telephone interview at 3 months to assess goals of care
  ACP video decision aid: 10 minute video decision aid describing the goals-of-care options
- Standard Care: * In-person interview where the patient and caregiver dyad will randomized to either the video aid intervention or standard care and complete baseline questionnaire
  * Receive the verbal description of the three types of care
  * Follow telephone interview at 3 months
  Usual Care: Verbal description of the three types of care
Arm/Group | ACP Video Decision Aid | Standard Care
Number analyzed (Participants) | 25 | 25
Participants
  Concordance in goals of care pre intervention: Number of dyads with concordant goals of care | 20 | 15
  Concordance in goals of care pre intervention: Number of dyads with disconcordant goals of care | 5 | 10
  Concordance in goals of care post intervention: Number of dyads with concordant goals of care | 13 | 15
  Concordance in goals of care post intervention: Number of dyads with disconcordant goals of care | 12 | 10
  Concordance in goals of care 3 months post intervention: Number of dyads with concordant goals of care | 10 | 9
  Concordance in goals of care 3 months post intervention: Number of dyads with disconcordant goals of care | 15 | 16

2. Secondary Outcome: Increased Advance Care Planning (ACP) Conversations
Description: Patients randomized to the video will have more ACP conversations and documentation after 3 months.
Time Frame: Baseline and 3 months
Population: AYA participants that had data at 3-month follow-up
Measure: Count of Participants; unit: Participants
Groups:
- Standard Care - Patient: The research study procedures include: screening for eligibility and study interventions including questionnaires and follow up visits.
  * In-person interview where the patient and caregiver together will randomized to either the video aid intervention or standard care
  * Receive the verbal description of the three types of care
  * Follow telephone interview at 3 months
  Usual Care-: Verbal description of the three types of care
Arm/Group | ACP Video Decision Aid - Patient | Standard Care - Patient
Number analyzed (Participants) | 23 | 22
Participants
  Change in number of AYAs that engaged in ACP conversations following the intervention to 3-months | 13 | 13
  Change in number of AYAs that had ACP documentation from baseline to 3 months | 2 | 4

ADVERSE EVENTS:
Time Frame: Through study completion; average of 3-months, ending 5/2022
Groups:
- Standard Care - Caregiver: The research study procedures include: screening for eligibility and study interventions including questionnaires and follow up visits.
  * In-person interview where the patient and caregiver together will randomized to either the video aid intervention or standard care
  * Receive the verbal description of the three types of care
  * Follow telephone interview at 3 months
  Usual Care-: Verbal description of the three types of care
Arm/Group | ACP Video Decision Aid - Patient | ACP Video Decision Aid - Caregiver | Standard Care - Patient | Standard Care - Caregiver
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 2/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/04/NCT04149704/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/04/NCT04149704/ICF_001.pdf